CLINICAL TRIAL: NCT00100529
Title: Stereo Photogrammetry Soft Tissue in Normal Individuals and Patients With Craniofacial Dysmorphologies
Brief Title: Stereo Photogrammetry Imaging in Normal Volunteers and Patients With Head and Facial Malformations
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050052; 05-D-0052
Record Dates: First submitted 2004-12-31; First posted 2005-01-03 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2012-06-29

CONDITIONS: Craniofacial Abnormalities
Keywords: Facial Imaging; Genetics; Growth; Development; Diagnostics; Craniofacial Dysmorphologies; Facial Features
MeSH Terms: conditions — Craniofacial Abnormalities

SUMMARY:
This study will use stereo photogrammetry to: 1) characterize facial features of genetic and congenital malformations; 2) define facial features associated with normal growth and development; and 3) determine if stereo photogrammetry soft tissue imaging can be used to help diagnose head and facial malformations. These abnormalities currently are diagnosed using 2- or 3-dimensional skeletal images obtained with x-rays. Stereo photogrammetry uses a camera and computer to generate 3-dimensional images of the soft tissues of the face. Because the method does not use any radiation, images can be taken repeatedly to evaluate patients over a long term.

Using stereo photogrammetry, images of people who belong to a defined group, for example, 17-year-old Caucasian males, can be combined (or morphed) into one image, allowing measurement of the facial features of the group. Comparing the morphed images of a normal control group with those of people with specific genetic conditions may reveal distinctions that could be used in diagnosing conditions that are currently diagnosed using x-rays.

Healthy normal volunteers and patients with craniofacial dysmorphologies may be eligible for this study. Patients are recruited from current NIH studies of various genetic diseases. People who have previously had head and neck surgeries, including cosmetic surgery, may not participate.

Participants give a medical and dental history, including any orthodontic work or facial surgeries. They are then positioned in front of a photogrammetry camera, a headband is placed on their head, and their picture is taken. A coded patient number is entered into the computer, where the image is stored until further analysis. Most participants are evaluated one time, but some patients and control subjects may be asked to return yearly for repeat images.

DETAILED DESCRIPTION:
In previous decades, analysis of craniofacial dysmorphologies have been conducted using two- or three-dimensional imaging of skeletal tissues acquired through radiography, with little analysis of soft tissue structures. The advantages of stereophotogrammetry surface scanning include easy image acquisition, the procedure is non-invasive, and images may be easily repeatedly taken for longitudinal evaluation of facial morphology. No radiation is used in acquiring these images.

The purposes of this study are to: 1) characterize the surface tissue facial features in different genetic diseases and syndromes; 2) define facial parameters of age-related growth and development; and 3) establish the use of stereophotogrammetry surface tissue imaging in aiding the diagnosis of genetic conditions and prediction of the clinic course of craniofacial dysmorphologies and associated genotypes.

Procedures will entail the acquisition of facial images from patients with known and suspected dysmorphologies as well as healthy controls. Facial parameters of various patient groups will be characterized in a standardized manner. In addition, composite (mean) images of patients with a particular diagnosis will be compared with controls using software algorithms. These facial parameters will be used to calculate the sensitivity and specificity of this technology to predict the genetic dysmorphology.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male and female subjects of all ages and racial groups. The lower age limit will be determined by the ability to cooperate with imaging.
  2. Patient populations recruited from current NIH Intramural Studies with various defined genetic diseases such as Fanconi anemia.
  3. Controls recruited from the families of patients with genetic or congenital diseases, healthy volunteers participating in other NIH studies, or non-affected populations at collaborating institutions.

EXCLUSION CRITERIA:

1. Patients or controls with a history of head and neck surgery to include cosmetic facial surgery.
2. Patients unable to cooperate with imaging.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1813 (Actual)
Dates: Start 2004-12-21; Study Completion 2012-06-29

CONTACTS AND LOCATIONS:
Overall Officials: Carol W Bassim, D.M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (3):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Associacao dos Gemeos do Norte de Minas Gerais, Minas Gerais, Brazil
- Universidad Peruana Cayetano Heredia, Lima, Peru

REFERENCES:
- [Background] Li Y, Shum HY, Tang CK, Szeliski R. Stereo reconstruction from multiperspective panoramas. IEEE Trans Pattern Anal Mach Intell. 2004 Jan;26(1):45-62. doi: 10.1109/tpami.2004.1261078. PMID 15382685
- [Background] Hart TC, Marazita ML, Wright JT. The impact of molecular genetics on oral health paradigms. Crit Rev Oral Biol Med. 2000;11(1):26-56. doi: 10.1177/10454411000110010201. PMID 10682900
- [Background] Szeliski R, Scharstein D. Sampling the disparity space image. IEEE Trans Pattern Anal Mach Intell. 2004 Mar;26(3):419-25. doi: 10.1109/TPAMI.2004.1262341. PMID 15376889